CLINICAL TRIAL: NCT05060341
Title: Long-Term Follow-Up Study of Participants Enrolled in the MGT016 Phase 1, Open-Label, Dose-Escalation Study of AAV2hAQP1 for Radiation-Induced Parotid Gland Hypofunction and Xerostomia
Brief Title: Long-Term Follow-Up Study of AAV2hAQP1 for Radiation Induced Xerostomia
Status: Active, not recruiting | Type: Observational
Sponsor: MeiraGTx, LLC (Industry)
Responsible Party: Sponsor
Organization: MeiraGTx UK II Ltd (Industry)
Other Study IDs: MGT-AQP1-102
Record Dates: First submitted 2021-03-09; First posted 2021-09-29 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Radiation-induced Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a long-term follow-up study for patients who have been administered AAV2hAQP1 in the Phase 1 Open-Label, Dose Escalation Study to Determine the Optimal Dose, Safety, and Activity in Subjects with Radiation Induced Parotid Gland Hypofunction and Xerostomia

DETAILED DESCRIPTION:
This clinical trial is designed to assess the long-term safety and activity of intra-parotid administration of AAV2hAQP1 in subjects with radiation-induced parotid salivary hypofunction and xerostomia.

After completion of their Month 12 Follow-Up visit in Study MGT016, subjects will be invited to enroll in this 4-year follow-up study during which they will be assessed for up to 60 months following study drug administration. This follow-up trial is a non-interventional study designed to collect data on longer-term safety and activity at 18, 24, 36, 48, and 60 months following study drug administration.

Over the course of the study, subjects will undergo physical and oral examinations; vital sign measurements; weight measurements; AE assessments; concurrent medication assessments; sample blood collection for hematology and chemistry; urinalysis; ear, nose, and throat (ENT) screening for malignancy; imaging assessments (if indicated); salivary flow assessments; and questionnaire assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Are willing and able to provide informed consent
2. Received AAV2hAQP1 administered via Stensen's duct to a single or both parotid glands in the prior open-label, Phase 1, dose-escalation study (Study MGT016)
3. Are willing and able to adhere to the protocol and long-term follow-up

Exclusion Criteria:

1. Subjects unwilling or unable to meet with the requirements of the study will be excluded

Ages: 18 Years to 81 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with radiation induced parotid gland hypofunction and xerostomia who have particpated in the MGT016 AAV2hAQP1 study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
• Incidence of AEs, treatment-emergent adverse events (TEAEs), and SAEs | 4 years
  Safety

SECONDARY OUTCOMES:
Changes in saliva flow compared to baseline. | 4 years
  Changes in unstimulated and stimulated salivary output (mL/minute) of the treated parotid gland and/or whole saliva output as compared to baseline.
Changes in the McMaster Global Rate of Change relative to Baseline | 4 years
  This first part of this questionnaire asks the patient to evaluate their Dry Mouth relative to before treatment as better, worse, or the same. If better or worse, the patient is asked to rate the magnitude of change, on a scale of 1-7, with a higher score being a better outcome.
  This first part of this questionnaire asks the patient to evaluate how limited they are in daily activities due to dry mouth, relative to before treatment as better, worse, or the same. If better or worse, the patient is asked to rate the magnitude of change, on a scale of 1-7, with a higher score being a better outcome.
Changes in the Xerostomia Questionnaire relative to Baseline | 4 years
  The XQ is a series of 8 questions designed to assess the degree of xerostomia symptoms. Each question is a scale of 1-10, with high values indicating worse xerostomia.
Changes in the MD Anderson Symptom Inventory - Head and Neck | 4 years
  The MDASI-HN is a questionnaire consisting of 28 questions designed to assess the degree of xerostomia symptoms. Each question is a scale of 1-10, with high values indicating worse xerostomia.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Leland Stanford Junior University, Stanford, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Atrium Health, Charlotte, North Carolina
- Health Sciences North - Northeast Cancer Center, Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No